CLINICAL TRIAL: NCT02632227
Title: Prediction of Fluid Responsiveness Using TFU (Transfontanel Ultrasound) in Children With Congenital Heart Disease After Cardiac Surgery
Brief Title: Fluid Responsiveness Using TFU (Transfontanel Ultrasound) in Children With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Other Study IDs: 1511-105-0724
Record Dates: First submitted 2015-12-13; First posted 2015-12-16 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Fluid Responsiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hypovolemia: patients with hypovolemic signs including hypotension, decreased central venous pressure (less than 5mmHg), and decreased urine output
  Interventions: Procedure: TFU(transfontanel ultrasound)

INTERVENTIONS:
Procedure: TFU(transfontanel ultrasound) — The respiratory variation of the carotid artery blood flow peak velocity was measured using TFU before and after the fluid administration (10ml/kg for 20 min.)

SUMMARY:
The purpose of this study was to evaluate the clinical usefulness of TFU (transfontanel ultrasound)for the prediction of fluid responsiveness in children undergoing congenital heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing cardiac surgery

Exclusion Criteria:

* preterm closure of anterior fontanelle
* anatomical abnormalities on aortic arch (ex, patent ductus arteriosus)
* presence of intracardiac and extracardiac shunt

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients with congenital heart disease undergoing cardiac surgery
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2017-03 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
change in respiratory variation of carotid artery blood flow peak velocity after volume expansion | before and after fluid administration (20min)

SECONDARY OUTCOMES:
change in cardiac index after volume expansion | before and after fluid administration (20min)
change in pleth variability index after volume expansion | before and after fluid administration (20min)
change in respiratory variation of aorta flow blood flow peak velocity after volume expansion | before and after fluid administration (20min)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea